CLINICAL TRIAL: NCT04690699
Title: LUMINOS-103: A Basket Trial Evaluating the Safety and Efficacy of Lerapolturev (PVSRIPO) and Lerapolturev in Combination With Anti-PD-1/L1 Checkpoint Inhibitors in Patients With Advanced Solid Tumors
Brief Title: LUMINOS-103: A Basket Trial of Safety & Efficacy of Lerapolturev With or Without Checkpoint Inhibitors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: business decision
Sponsor: Istari Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUMINOS-103
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor; Bladder Cancer; Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — DDMS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort E: Lerapolturev (Experimental): Subjects will be treated with lerapolturev by intravesical instillation
  Interventions: Biological: Lerapolturev
- Cohort F: Lerapolturev + 5% DDM (Experimental): Subjects will be treated with lerapolturev by intravesical instillation after a sequence of 5% DDM and saline washes
  Interventions: Biological: Lerapolturev; Other: 5% DDM

INTERVENTIONS:
Biological: Lerapolturev — Lerapolturev administered via intravesical instillation once
Other: 5% DDM — 5% DDM and saline washes
  Arms: Cohort F: Lerapolturev + 5% DDM

SUMMARY:
This is a Phase 1/2, open-label, multi-center, single arm basket study evaluating the administration of lerapolturev ± anti programmed cell death protein 1 (PD 1)/programmed death-ligand 1 (PD L1) monoclonal antibody (mAb) (which will be referred to throughout this protocol as "anti-PD-1/L1 therapy") therapy in adult patients with solid tumor cancers. Non-muscle invasive Bladder Cancer has been selected as the tumor specific cancer of interest for enrollment.

DETAILED DESCRIPTION:
Patients with recurrent non-muscle invasive bladder cancer (NMIBC) intended for transurethral resection of bladder tumor (TURBT) or cystectomy will receive lerapolturev by intravesical instillation. Approximately 12-15 patients will be enrolled.

ELIGIBILITY:
Master Protocol Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Age ≥ 18 years of age at the time of signing the informed consent.
3. Prior CDC-recommended vaccination series against PV and has received a boost immunization with trivalent Poliovirus Vaccine Inactivated (IPOL®) (Sanofi-Pasteur SA) at least 1 week, but less than 6 weeks, prior to Cycle 1 Day 1.

   * Note: Patients who are unsure of their vaccination status must provide evidence of anti-PV immunity prior to enrollment, as applicable.
4. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
5. A formalin-fixed paraffin-embedded (FFPE) tumor specimen (from archival or fresh biopsy) with an associated pathology report documenting the histology of the tumor type of interest must be confirmed to be available to send to the Sponsor.

   * Note: additional details can be found in the tumor specific appendix.
6. Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
7. Adequate bone marrow and liver function as assessed by the following:

   * Hemoglobin ≥9.0 g/dl (patients may be transfused)
   * Lymphocyte count ≥ 0.5 x 109/L (500/µL)
   * Absolute neutrophil count (ANC) ≥1.5 x 109/L (1500/µL)
   * Platelet count ≥100 x 109/L (100,000/µL) without transfusion
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)

     * Subjects with documented liver metastases: AST and ALT ≤5 x ULN
   * Serum total bilirubin ≤1.5 x ULN OR direct bilirubin <ULN for patients with total bilirubin > 1.5 x ULN
   * For patients not receiving therapeutic anticoagulation: international normalized ratio (INR), prothrombin time (PT), partial thromboplastin time (PTT) (or activated partial thromboplastin time [aPTT]) ≤ 1.5 x ULN
8. Resolution of nonhematologic toxicities from prior therapy or surgical procedures to

   ≤ Grade 1 or baseline (except alopecia).
9. Contraceptive use by men or women of childbearing potential should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Master Protocol Exclusion Criteria:

1. Any radiotherapy, chemotherapy, immunotherapy, biological, investigational, or hormonal therapy for cancer treatment (except for adjuvant hormonal therapy for breast cancer or prostate cancer defined as M0 disease or prostate-specific antigen persistence/recurrence without metastatic disease) within 21 days of Cycle 1 Day 1.
2. Patients requiring anticoagulation with warfarin are excluded. Additional eligibility criteria for anticoagulation requirements for each solid tumor cancer of interest will be provided in the tumor specific appendix.
3. Presence of central nervous system (CNS) metastases requiring immediate treatment with radiation therapy or steroids (ie, patient must be off steroids administered for brain metastases for ≥ 14 days prior to Cycle Day 1). Leptomeningeal disease is excluded regardless of clinical stability or treatment status.
4. Clinically significant (ie, active) cardiovascular disease at the time of signing the informed consent; for example, cerebrovascular accidents (≤ 6 months before the first dose of lerapolturev, myocardial infarction (≤ 6 months before the first dose of lerapolturev), unstable angina, serious cardiac arrythmia requiring medication, or uncontrolled symptomatic congestive heart failure [Class II or higher as defined by the New York Heart Association [NYHA] functional classification system; see Appendix 4]).
5. QTcF interval > 450 msec (males) or > 470 msec (females) at Screening (confirmed in triplicate). For patients with ventricular pacemakers or bundle branch block, QTcF >500 msec.
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Cycle Day 1, or anticipation of the need for major surgical procedure during the course of the study.
7. Active or history of autoimmune disease or immune deficiency within previous 2 years, with the following exceptions:

   * History of autoimmune-related hypothyroidism that is managed by thyroid replacement hormone
   * Type 1 diabetes mellitus that is well-controlled (as determined by the Investigator) by an established insulin regimen
   * Eczema, psoriasis, or lichen simplex chronicus with dermatologic manifestations only (eg, patients with psoriatic arthritis are excluded), provided all of the following conditions are met:

     * Rash must cover < 10% of body surface area
     * Disease is well-controlled (as determined by the Investigator) at baseline and requires only low-potency topical corticosteroids
     * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within 12 months of Cycle 1 Day 1
8. History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

   * History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
9. Uncontrolled pleural effusion, pericardial effusion, or ascites; patients with indwelling catheters (eg, PleurX®) are allowed.
10. Known serious active infection (eg, human immunodeficiency virus [HIV], hepatitis B or C, tuberculosis, etc.).

    * Participants with a negative hepatitis B surface antigen (HBsAg) test and a positive total hepatitis B core antibody (HBcAb) test are allowed.
    * History of positive hepatitis C virus (HCV) antibody test, but negative HCV RNA test is allowed.
    * Participants with a historical positive HIV test are not allowed.
11. Treatment with systemic immunosuppressive medication within 28 days of Cycle 1 Day 1, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (eg, 48 hours of corticosteroids for a contrast allergy) are eligible.
    * Patients receiving mineralocorticoids (eg, fludrocortisone), or systemic prednisone equivalent corticosteroid doses of < 10 mg per day are eligible for the study.
12. Prior allogeneic or autologous hematopoietic stem cell or bone marrow transplantation.
13. Receipt of any live, attenuated vaccines within 28 days of Cycle 1 Day 1. Vaccination to prevent symptomatic SARS-CoV-2 infection is allowed as long as the vaccine is NOT a live attenuated vaccine (e.g. adenovirus-based constructs); however, the vaccine should be administered ≥ 1 week before or after a lerapolturev injection.
14. Known hypersensitivity to any of the drugs used in this study.
15. Pregnant or lactating women.
16. History of human serum albumin allergy.
17. History of neurological complications due to PV infection.
18. History of agammaglobulinemia.
19. Legal incapacity or limited legal capacity.
20. Other uncontrolled serious chronic disease or psychiatric condition that in the Investigator's opinion could affect the patient's safety, compliance, or follow-up in the protocol.

Non-Muscle Invasive Bladder Cancer Specific Inclusion Criteria:

1. Prior history of stage Ta, T1, or Tis urothelial carcinoma of the bladder

   1. Tumors with up to 50% squamous or glandular differentiation are eligible
   2. History of variant bladder histologies are excluded (eg, sarcomatoid, plasmacytoid, small cell or neuroendocrine, pure pure squamous cell carcinoma, pureadenocarcinoma, micropapillary, nested, lymphepithelioma-like, clear cell)
2. Documented tumor recurrence at cystoscopy where the tumor is amenable to TURBT or cystectomy.
3. Measured or calculated (per institutional standard) creatinine clearance ≥ 45 ml/min (glomerular filtration rate [GFR] can also be used in place of creatinine clearance).
4. If the patient has an available formalin-fixed paraffin-embedded (FFPE) tumor specimen with an associated pathology report documenting NMIBC, the specimen must be confirmed to be available to send to the Sponsor. Patients without an available FFPE specimen are still eligible to enroll.
5. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 is NOT required. This is an exception to the inclusion criterion outlined in the master protocol.

Non-Muscle Invasive Bladder Cancer Specific Exclusion Criteria:

1. Patients with exposure to intravesical agents (e.g. BCG, mitomycin C, epirubicin, oncolytic viruses, anti-PD-1/L1 inhibitors, investigational therapies, etc.) within 3 months prior to the administration of lerapolturev.
2. Patients whose anticoagulation or antiplatelet medications cannot be managed by local institutional guidelines to accommodate the safe intravesical instillation of lerapolturev followed by TURBT, as determined by the treating physician.
3. Received prior radiation to the pelvis.
4. Received prior systemic therapy for bladder cancer, including PD-1/L1 inhibitors.
5. History of vesicoureteric reflux or an indwelling urinary stent.
6. History of stage T2 or higher bladder cancer
7. Medical conditions (as determined by the investigator) that would interfere with the ability of the patient to retain urine for 2 hours. Examples include urinary incontinence, overactive bladder, or low bladder compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Franklin, Study Director — Istari Oncology
Locations (1):
- Carolina Urologic Research Center, Myrtle Beach, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort E: Lerapolturev | Cohort F: Lerapolturev + 5% DDM
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study closed prior to reaching enrollment goal due to business decision.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort E: Lerapolturev | Cohort F: Lerapolturev + 5% DDM | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 75.5 [65 to 87] |  | 75.5 [65 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 4 |  | 4
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Underwent TURBT or Cystectomy as Scheduled
Description: To evaluate the safety and tolerability of lerapolturev monotherapy administered by intravesical instillation to patients with recurrent NMIBC intended for TURBT or cystectomy
Time Frame: 1 month
Population: Study closed prior to meeting enrollment goal due to business decision
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort E: Lerapolturev | Cohort F: Lerapolturev + 5% DDM
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days post-dose
Description: AE were determined by investigator assessment, laboratory evaluation, and patient self-reporting. All AE were graded per NCI CTCAE v5.
Arm/Group | Cohort E: Lerapolturev | Cohort F: Lerapolturev + 5% DDM
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort E: Lerapolturev (N=4) | Cohort F: Lerapolturev + 5% DDM (N=0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04690699/Prot_SAP_000.pdf